CLINICAL TRIAL: NCT01702844
Title: LCCC 1210 - Phase II, Multicenter, Single Arm Study of the Tolerability of Weekly Nab-paclitaxel as Second Line Treatment for Elderly Patients With Advanced Lung Cancer
Brief Title: Single Arm on the Tolerability of Weekly Nab-paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1210
Record Dates: First submitted 2012-09-25; First posted 2012-10-08 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: Nab paclitaxel; Abraxane; First Line; Non small cell lung cancer; NSCLC; Phase II; Non-Randomized; Elderly; Lineberger; UNC; LCCC 1210
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab paclitaxel (Experimental): Patients will receive nab-paclitaxel once weekly for 3 weeks of every 4 week cycle
  Interventions: Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Nab-Paclitaxel — Administer 2 cycles of Nab-Paclitaxel 100 mg/m2 IV on days 1 8 and 15
  Other Names: Abraxane

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of weekly nab-paclitaxel for a second-line treatment in elderly subjects, 70 years of age or greater, with non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This will be a non-randomized phase II study evaluating the safety and efficacy of weekly nab-paclitaxel for second-line treatment in 42 elderly patients, who are 70 years of age or greater with non-small cell lung cancer (NSLC). Patients will be required to have progressed on a single prior regimen. Nab-paclitaxel 100mg/m2 will be administered intravenously, weekly for 3 weeks of every 4-week cycle. After every two cycles of therapy, imaging will be performed to assess for response. Patients will be eligible to continue receiving therapy until the time of disease progression.

Primary Objectives To evaluate the tolerability of weekly nab-paclitaxel in older adults with advanced lung cancer who have progressed on at least 1 prior regimen after 6 cycles or 3 weeks after discontinuation of treatment, for those who come off treatment earlier.

Secondary Objectives To estimate overall survival To estimate progression-free survival To estimate the response rate

Correlative Objectives To explore baseline components of the Geriatric Assessment (GA) as predictors of chemotherapy tolerance and overall survival To explore the use of p16 measurements in the elderly as predictors of chemotherapy tolerance and overall survival To explore the impact of weekly nab-paclitaxel treatment on quality of life, as measured by Lung Cancer Symptom Scale (LCSS) and Functional Assessment of Cancer Therapy-Lung (FACT-L).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female patient
* Greater than or equal to 70 years of age
* Diagnosis of NSCLC histologically or cytologically confirmed
* Internal Association for the Study of Lung Cancer Version 7 Stage IV disease or recurrence after prior surgery or radiotherapy
* Progression following one line of prior chemotherapy consisting of a platinum agent plus a standard cytotoxic partner agent other than a taxane, typically pemetrexed gemcitabine or vinorelbine
* A single agent non cytoxic regimen if the patient has a molecular change that the non cytotoxic regimen would be expected to be efficacious for epidermal growth factor receptor (EGFR) mutation for erlotinib and (EML4) anaplastic lymphoma kinase (ALk) or ROS1 for crizotinib
* Eastern Cooperative Oncology Group performance status 0 to 2
* Adequate organ and bone marrow function as defined by
* Absolute neutrophil count greater than or equal to 1500 cells/mm3
* Creatinine less than or equal to 1.5 mg dL
* Total bilirubin less than or equal to 1.5 mg dL
* Alkaline phosphatase less than or equal to 2.5 x upper limit of normal
* Alanine aminotransferase less than or equal to 2.5 x upper limit of normal
* Aspartate aminotransferase less than or equal to 2.5 upper limit of normal
* Recovered from all reversible toxicities related to their previous treatment to less than or equal to grade 1 or baseline
* Patients must have equal to grade 2 pre existing peripheral neuropathy
* Women of childbearing potential and sexually active men must agree to use effective contraception prior to study entry for the duration of study participation and for three months after completing treatment. Adequate contraception is defined as any medically recommended method as per standard of care
* Negative serum or urine bhCG pregnancy test at screening for patients of childbearing potential
* Patients with brain metastases may participate if they have undergone appropriate treatment for the lesions are at least two weeks post treatment without evidence for post treatment progression have no significant neurologic symptoms and no longer require steroids for the reason of brain metastases. Patients with symptoms suggestive of central nervous system (CNS) metastases should be evaluated with imaging prior to study participation

Exclusion Criteria:

* Prior taxane therapy for any indication
* Less than 3 weeks elapsed since prior exposure to chemotherapy
* Pre existing neuropathy greater than grade 1
* Other active invasive malignancy requiring ongoing therapy or expected to require systemic therapy within two years localized squamous cell carcinoma of the skin basal cell carcinoma of the skin, carcinoma in situ of teh cervix or other malignancies requiring locally ablative therapy only will not result in exclusion
* Concomitant anticancer therapy immunotherapy or radiation therapy within prior 4 weeks
* Have received treatment within the last 30 days prior to study entry with any drug that has not receive regulatory approval for an indication at the time of study entry
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection requiring IV antibiotics symptomatic congestive heart failure unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situations that would limit compliance with study requirements
* Pregnant women are excluded due to the potential for teratogenic or abortifacient effects of nab paclitaxel because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued prior to participation of the mother on study
* Known hypersensitivity to protein bound paclitaxel
* Any other concurrent condition that in the investigators opinion would jeopardize compliance with the protocol

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (8):
- United States (8):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Bon Secours Virginia Health System, Midlothian, Virginia
  - Swedish Cancer Institute, Seattle, Washington

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center homepage — http://unclineberger.org/
- See also: National Cancer Institute (NCI) homepage — http://www.cancer.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 participants were accrued between June 2013 and April 2017 at 7 institutions in the United States
Pre-assignment Details: Another 9 participants signed consent but did not start the trial due to screen failure (6), progression of disease prior to study start (1) and withdrawal of consent prior to start (2.)
Period: Overall Study
Arm/Group | Nab Paclitaxel
Started | 42
Disease Progression | 23
Completed | 23
Not Completed | 19
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | Nab Paclitaxel
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years] | 76.3 [71 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42
Smoking status [Count of Participants; unit: Participants]
  Never smoker | 4
  Former/current smoker | 38
Performance status [Count of Participants; unit: Participants] — East Coast Oncology Group (ECOG) Performance status: scale from 0-5 to describe a patient's level of functioning in terms of selfcare ability and activity level.
  0-Fully active
  1. Restricted in strenuous activity but ambulatory and able to carry out light work
  2. Ambulatory and capable of all selfcare but unable to carry out any work; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0, Fully active | 5
    1, Restricted in strenuous activity but ambulatory | 28
    2, limited selfcare | 9
Exercise [Count of Participants; unit: Participants] — Number of times participant exercises for at least 10 minutes per day
  Participants
    Never | 10
    Few times per month | 3
    1-2 times per week | 6
    3-4 times per week | 2
    More than or equal to 5 times per week | 1
    Unknown/Not reported | 20
Alcohol [Count of Participants; unit: Participants] — Participant report of whether or not they drink alcohol
  Participants
    No | 13
    Yes | 7
    Almost never | 7
    Unknown/Not reported | 15
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 35
  Squamous cell carcinoma | 7
Prior treatment regimens [Count of Participants; unit: Participants] — Prior cancer treatment regimens; participants could have more than one prior regimen
  Participants
    Carboplatin plus pemetrexed | 26
    Carboplatin, pemetrexed, and bevacizumab | 4
    Cisplatin plus pemetrexed | 1
    Carboplatin plus gemcitabine | 11
    Nivolumab | 8
    Erlotinib | 1
    Other prior regimens | 3
Best response to prior therapies [Count of Participants; unit: Participants]
  Complete response | 0
  Partial response | 3
  Stable disease | 16
  Progressive disease | 22
  Unknown/Not evaluable | 13
Frailty index [Count of Participants; unit: Participants] — Carolina Frailty Index (CFI) was derived from a cancer-specific geriatric assessment tool assessing functional status, comorbidity, psychological state, social support, nutritional support, medications, and cognition. CFI scores (range, 0-1) are categorized as robust (0-0.2), pre-frail (0.2-0.35), and frail (>0.35).
  Participants
    Robust (0 to <0.2) | 5
    Prefrail (0.2-0.35) | 10
    Frail (>0.35) | 11
    Unknown/Not assessed | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Without Any Adverse Events Grade 3 or Higher
Description: Tolerability of weekly nab-paclitaxel, as measured by occurrence of Grade 3 or worse toxicity after 6 cycles or 3 weeks after discontinuation of treatment, for those who came off treatment earlier as measured by the NCI Common Terminology Criteria for Adverse Events CTCAE, version 4. The CTCAE is a descriptive terminology utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 168 days after start of treatment (6 cycles) (or 3 weeks after discontinuation of treatment, for those who come off treatment earlier)
Measure: Count of Participants; unit: Participants
Arm/Group | Nab Paclitaxel
Number analyzed (Participants) | 42
Participants | 28

2. Secondary Outcome: Median Overall Survival
Description: Overall Survival is defined as the time from day 1 (D1) of treatment until death as a result of any cause
Time Frame: up to 2 years after end of treatment (treatment lasts up to 168 days (up to 6 cycles of 28 days each))
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nab Paclitaxel
Number analyzed (Participants) | 42
Months | 9.3 [6.4 to 12.1]

3. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival is defined as the time from D1 of treatment until progression or death as a result of any cause. Progressive Disease (PD) is determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. PD is at least a 20% increase in the sum of the longest diameters (LD) of the target lesions taking as reference the smallest sum LD recorded since the treatment started including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters. The appearance of one or more new lesions also constitutes PD.
Time Frame: up to 2 years after end of treatment (treatment lasts up to 168 days (up to 6 cycles of 28 days each))
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nab Paclitaxel
Number analyzed (Participants) | 42
Months | 5.2 [2.0 to 7.4]

4. Secondary Outcome: Overall Response Rate
Description: Response will be measured by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) version 1.1, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. The Overall Response rate is defined as the percentage of participants with CR or PR
Time Frame: as for outcome 1
Population: 4 subjects were not analyzed for this outcome due to lack of follow up disease assessments (off treatment after only one cycle for hospice and/or death)
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | Nab Paclitaxel
Number analyzed (Participants) | 38
percentage of patients with response | 34.2 [19.6 to 51.4]

ADVERSE EVENTS:
Time Frame: From day 1 of study treatment to 30 days after treatment is discontinued (with an average treatment duration of 168 days)
Arm/Group | Nab Paclitaxel
All-Cause Mortality (participants affected / at risk) | 41/42
Serious Adverse Events (participants affected / at risk) | 15/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab Paclitaxel (N=42)
Acute kidney injury (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Bronchial infection (Infections and infestations) | 1
Chills (General disorders) | 1
Confusion (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fever (General disorders) | 1
Gait disturbance (General disorders) | 1
Heart failure (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Stroke (Nervous system disorders) | 1
Vasculitis (Vascular disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab Paclitaxel (N=42)
Abdominal pain (Gastrointestinal disorders) | 5
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase i (Investigations) | 1
Alkaline phosphatase incre (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 12
Anal hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 18
Anorexia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase (Investigations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood and lymphatic system (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bronchial infection (Infections and infestations) | 2
Cardiac disorders - Other, (Cardiac disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine increased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 3
Dry mouth (Gastrointestinal disorders) | 2
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Edema limbs (General disorders) | 16
Endocrine disorders - Othe (Endocrine disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Eye disorders - Other, spe (Eye disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 26
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
General disorders and admi (General disorders) | 1
Generalized muscle weaknes (Musculoskeletal and connective tissue disorders) | 3
Genital edema (Reproductive system and breast disorders) | 1
Headache (Nervous system disorders) | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infusion site extravasatio (General disorders) | 1
Insomnia (Psychiatric disorders) | 2
Lymphocyte count decreased (Investigations) | 8
Metabolism and nutrition d (Metabolism and nutrition disorders) | 1
Mucosal infection (Infections and infestations) | 5
Mucositis oral (Gastrointestinal disorders) | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nail infection (Infections and infestations) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 12
Neutrophil count decreased (Investigations) | 15
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 2
Paronychia (Infections and infestations) | 2
Peripheral motor neuropath (Nervous system disorders) | 4
Peripheral sensory neuropa (Nervous system disorders) | 20
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Renal and urinary disorder (Renal and urinary disorders) | 1
Respiratory, thoracic and (Respiratory, thoracic and mediastinal disorders) | 1
Retinal vascular disorder (Eye disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Sinusitis (Infections and infestations) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 4
Supraventricular tachycard (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Transient ischemic attacks (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Upper respiratory infectio (Infections and infestations) | 6
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Vasculitis (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Watering eyes (Eye disorders) | 2
Weight gain (Investigations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT01702844/Prot_SAP_000.pdf